CLINICAL TRIAL: NCT03296566
Title: The SAFE Study: Satisfaction and Adherence to Follow-Up With Colposcopy Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other); Women's Health Research Institute of British Columbia (Other)
Responsible Party: Principal Investigator, Marette Lee, Program Director, BC Provincial Colposcopy Program, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H16-03194
Record Dates: First submitted 2017-07-20; First posted 2017-09-28 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Uterine Cervical Dysplasia; Uterine Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Liaison Intervention (Experimental): The participants randomized to the intervention group will be exposed to the patient liaison in receiving their colposcopy report results and recommendations. Rather than receive results from their referring/family physician, an experienced colposcopy nurse will contact participants once the colposcopists complete the final colposcopy report. The colposcopy nurse will provide an explanation of the colposcopy results and subsequent follow-up or treatment recommendations, be available to answer patient questions (within her scope), offer educational or support resources to patients.
  Interventions: Behavioral: Patient Liaison
- Control (No Intervention): The control group will receive the standard of care for colposcopy results reporting via their referring physician. Following their colposcopy visit, control patients are given a slip of paper reminding them to call their family/referring physician for their colposcopy results in three weeks if they have not yet been contacted. Upon receipt of the final pathology, colposcopy reports are prepared by the colposcopists and forwarded to family/referring physicians typically within 2-3 weeks of the visit. Patients then receive the results of their colposcopy report from their family/referring physician by whatever method of communication preferred by that provider.

INTERVENTIONS:
Behavioral: Patient Liaison — An experienced colposcopy nurse will contact participants once the colposcopists complete the final colposcopy report. The colposcopy report will inform the referring provider that these patients will be informed of the results. The colposcopy nurse will provide an explanation of the colposcopy results and subsequent follow-up or treatment recommendations, be available to answer patient questions (within her scope), offer educational or support resources to patients. She will forward any patient questions beyond her scope to the patient's colposcopist who may then provide answers to the patient liaison or to the patient directly depending on the complexity and nature of the question.
  Arms: Patient Liaison Intervention

SUMMARY:
This study is intended to improve the patient experience of communication of colposcopy results and follow-up recommendations to patients. Current practice involves results being forwarded from the colposcopy clinic to the family or referring physician who then informs the patient. We are testing an intervention informed by focus groups in which a trained colposcopy nurse (patient liaison) directly contacts patients with their results and follow-up recommendations while providing education and support. We will examine whether this intervention improves patient satisfaction, reduces anxiety, and improves rates of adherence to follow-up and treatment appointments compared to the current practice.

DETAILED DESCRIPTION:
Cervical cancer is the second most commonly diagnosed cancer and third leading cause of cancer death in women worldwide. Pre-cancerous cells can be detected with regular Pap smear screening and diagnosed and treated with colposcopy. This process is limited by patient adherence to the follow-up and treatment recommendations. Currently at Vancouver General Hospital (VGH), the largest colposcopy clinic in the province, results are forwarded from the colposcopy clinic to the family or referring physician who informs patients of results and recommendations. Inefficiencies or errors in this step may cause patient dissatisfaction, missed appointments, increased costs, and compromise patient outcomes. The primary objective of this study is to examine whether having a trained colposcopy nurse directly contact patients with their results and follow-up recommendations while providing education and support will improve patient satisfaction and reduce anxiety, with the secondary aim being to assess the clinical effectiveness of this intervention in improving rates of adherence to follow-up and treatment appointments and potentially long-term clinical outcomes. The first phase of the study involves patient focus groups that will be interviewed about what elements of a patient liaison interaction are most important (separate Ethics submission). This information will inform the development of the patient liaison role and approaches to patient interaction to be utilized in the intervention in the second phase. The second phase will entail a randomized controlled trial comparing patient anxiety, satisfaction and adherence to follow-up between a control group (current practice) versus the intervention group exposed to the patient liaison at the VGH Colposcopy Clinic. For the primary aim, a questionnaire containing items pertaining to patient anxiety and satisfaction with their experience of receiving their colposcopy results will be administered both to the intervention and control groups and the mean scores pertaining to anxiety and satisfaction will be compared using two-tailed t-tests. For the secondary aim, a chart review at 6-12 months following the initial colposcopy visit will examine the rates of compliance with the recommended follow-up or treatment visits and histologic diagnoses, and comparisons will be sought between the intervention and control groups using z-score test.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 19 years of age or older
2. Must be patients presenting for an initial visit at the VGH Colposcopy Clinic

Exclusion Criteria:

1. Inability to speak conversational English- required to complete the questionnaire as well as provide informed consent to participate
2. Inability or refusal to provide consent
3. Pregnant - pregnant women do not usually have biopsies and their subsequent care may be much different than non-pregnant patients
4. Do not have a family physician or referring physician who will provide continuity of care following colposcopy - these patients do not have the option of getting results from a family or referring physician, so they would bias results.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marette Lee, MD/MPH/FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasubramani L, Orbell S, Hagger M, Brown V, Tidy J. Can default rates in colposcopy really be reduced? BJOG. 2008 Feb;115(3):403-8. doi: 10.1111/j.1471-0528.2007.01594.x. PMID 18190379
- [Background] Boone JD, Erickson BK, Huh WK. New insights into cervical cancer screening. J Gynecol Oncol. 2012 Oct;23(4):282-7. doi: 10.3802/jgo.2012.23.4.282. Epub 2012 Sep 19. PMID 23094132
- [Background] Bredart A, Kop JL, Efficace F, Beaudeau A, Brito T, Dolbeault S, Aaronson N; EORTC Quality of Life Group. Quality of care in the oncology outpatient setting from patients' perspective: a systematic review of questionnaires' content and psychometric performance. Psychooncology. 2015 Apr;24(4):382-94. doi: 10.1002/pon.3661. Epub 2014 Sep 5. PMID 25196048
- [Background] Byrom J, Clarke T, Neale J, Dunn PD, Hughes GM, Redman CW, Pitts M. Can pre-colposcopy sessions reduce anxiety at the time of colposcopy? A prospective randomised study. J Obstet Gynaecol. 2002 Jul;22(4):415-20. doi: 10.1080/01443610220141407. PMID 12521468
- [Background] Dietrich AJ, Tobin JN, Cassells A, Robinson CM, Greene MA, Sox CH, Beach ML, DuHamel KN, Younge RG. Telephone care management to improve cancer screening among low-income women: a randomized, controlled trial. Ann Intern Med. 2006 Apr 18;144(8):563-71. doi: 10.7326/0003-4819-144-8-200604180-00006. PMID 16618953
- [Background] Lerman C, Hanjani P, Caputo C, Miller S, Delmoor E, Nolte S, Engstrom P. Telephone counseling improves adherence to colposcopy among lower-income minority women. J Clin Oncol. 1992 Feb;10(2):330-3. doi: 10.1200/JCO.1992.10.2.330. PMID 1732434
- [Background] Litchfield IJ, Bentham LM, Lilford RJ, McManus RJ, Greenfield SM. Patient perspectives on test result communication in primary care: a qualitative study. Br J Gen Pract. 2015 Mar;65(632):e133-40. doi: 10.3399/bjgp15X683929. PMID 25733434
- [Background] Nugent LS, Tamlyn-Leaman K, Isa N, Reardon E, Crumley J. Anxiety and the colposcopy experience. Clin Nurs Res. 1993 Aug;2(3):267-77. doi: 10.1177/105477389300200304. PMID 8401241
- [Background] O'Connor M, Gallagher P, Waller J, Martin CM, O'Leary JJ, Sharp L; Irish Cervical Screening Research Consortium (CERVIVA). Adverse psychological outcomes following colposcopy and related procedures: a systematic review. BJOG. 2016 Jan;123(1):24-38. doi: 10.1111/1471-0528.13462. Epub 2015 Jun 22. PMID 26099164
- [Background] Percac-Lima S, Ashburner JM, Zai AH, Chang Y, Oo SA, Guimaraes E, Atlas SJ. Patient Navigation for Comprehensive Cancer Screening in High-Risk Patients Using a Population-Based Health Information Technology System: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jul 1;176(7):930-7. doi: 10.1001/jamainternmed.2016.0841. PMID 27273602
- [Background] Towler BP, Irwig LM, Shelley JM. The adequacy of management of women with CIN 2 and CIN 3 Pap smear abnormalities. Med J Aust. 1993 Oct 18;159(8):523, 526-8. PMID 8412951

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 297 participants were recruited and subsequently randomized. Post-randomization, 3 participants withdrew from the control arm. 294 patients were analyzed in the statistical analysis.
Groups:
- Patient Liaison Intervention: The participants randomized to the intervention group will be exposed to the patient liaison in receiving their colposcopy report results and recommendations. Rather than receive results from their referring physician, an experienced colposcopy nurse will contact participants once the colposcopists complete the final colposcopy report.
  Patient Liaison: An experienced colposcopy nurse will contact participants once the colposcopists complete the final colposcopy report. The colposcopy report will inform the referring provider that these patients will be informed of the results. The colposcopy nurse will provide an explanation of the colposcopy results and subsequent follow-up or treatment recommendations, be available to answer patient questions (within her scope), offer educational or support resources to patients. She will forward any patient questions beyond her scope to the patient's colposcopist.
Period: Overall Study
Arm/Group | Patient Liaison Intervention | Control
Started | 145 | 152
Completed | 126 | 103
Not Completed | 19 | 49
Not completed — Lost to Follow-up | 19 | 46
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: 297 consenting women >18 years old presenting for initial appointment at the study colposcopy clinic were randomized.
  Although 152 participants were randomized to the control group, 3 withdrew post-randomization and only 149 were included in the analysis (thus, a total of 294 participants were included in the analysis).
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Liaison Intervention | Control | Total
Number analyzed (Participants) | 145 | 149 | 294
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [28 to 43.5] | 31 [27 to 44] | 33 [27 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 149 | 294
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 111 | 90 | 201
  Unknown or Not Reported | 29 | 55 | 84

OUTCOME MEASURES:

1. Primary Outcome: Anxiety
Description: Mean state anxiety scores as measured by the State Trait Anxiety Inventory (STAI) State Subscale. The STAI has 40 items with 20 items allocated to each of the State Anxiety and Trait Anxiety subscales. Responses for the State Anxiety scale assess intensity of current feelings from 1-4 "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Item scores are added to obtain subtest total scores and for anxiety-present items, a higher score suggests higher anxiety. Scoring is reversed for anxiety-absent items (items in which a higher score suggests lower anxiety). Range of scores for the subscale is 20-80 with a higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the State Anxiety scale.
Time Frame: To be collected by questionnaire in 4-6 weeks following colposcopy visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Liaison Intervention | Control
Number analyzed (Participants) | 126 | 103
score on a scale | 37.3 (12.8) | 40.7 (11.2)

2. Primary Outcome: Quantitative Satisfaction With Colposcopy Visit Experience Including Interactions With Colposcopy Professionals
Description: Patient satisfaction scores as measured by items in the questionnaire drawn from the Visit Specific Satisfaction Instrument (VSQ-9) Inventory. The VSQ-9 is a 9 item survey that measures patient satisfaction with access to primary care, with the direct interaction with the physician, and with the visit overall on a scale ranging from 1 (poor) to 5 (excellent). To score the VSQ-9, responses from each individual are transformed linearly to a 0 to 100 scale, with 100 corresponding to "excellent" and 0 corresponding to "poor" (0= Poor, 25= Fair, 50= Good, 75= Very Good, 100= Excellent). The 9 responses are then averaged together to create a VSQ-9 overall score for each person, again with 100 being the best evaluation and 0 the poorest.
Time Frame: To be collected by questionnaire in 4-6 weeks following colposcopy visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Liaison Intervention | Control
Number analyzed (Participants) | 126 | 103
score on a scale | 68.3 (19.2) | 66.6 (18.2)

3. Primary Outcome: Satisfaction With Colposcopy Information and Diagnosis Education
Description: Satisfaction with information and education received regarding colposcopy, patient diagnosis and follow-up recommendations measured by questionnaire items that measure these factors (PSQ-18 Inventory). This inventory contains 18 items assessing each of the 7 dimensions of satisfaction with medical care (general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with doctor, accessibility and convenience). Each item is scored from 1-5. Some PSQ-18 items are worded so that agreement reflects satisfaction with medical care, whereas other items are worded so that agreement reflects dissatisfaction with medical care. All items all scored so that high scores reflect satisfaction with medical care. All items are then summed; sum score of all items may range from 18 to 90 points, where 18 points is the poorest evaluation and 90 points the best.
Time Frame: To be collected by questionnaire in 4-6 weeks following colposcopy visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Liaison Intervention | Control
Number analyzed (Participants) | 126 | 103
score on a scale | 65.6 (11.4) | 65.1 (11.1)

4. Secondary Outcome: Patient Knowledge of Own Colposcopy Diagnosis
Description: The percent of patients who correctly report their colposcopy pathologic diagnosis
Time Frame: To be collected by questionnaire in 4-6 weeks following colposcopy visit
Measure: Number; unit: percentage of participants
Arm/Group | Patient Liaison Intervention | Control
Number analyzed (Participants) | 126 | 103
percentage of participants | 66.3 | 84

5. Secondary Outcome: Adherence to Colposcopy Treatment and Follow-up Instructions
Description: Percentage of patients who attended follow-up at the colposcopy clinic
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Patient Liaison Intervention | Control
Number analyzed (Participants) | 126 | 103
percentage of participants | 61.4 | 52.3

ADVERSE EVENTS:
Time Frame: 6 months following recruitment
Description: The intervention is delivery of colposcopy results. The highest risk serious adverse event (with associated mortality risk) would be failure of colposcopy results delivery leading to failure to receive treatment for cervical dysplasia or carcinoma which may lead to a delay or absence of appropriate treatment with associated morbidity or mortality.
Arm/Group | Patient Liaison Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/149
Other Adverse Events (participants affected / at risk) | 0/145 | 0/149

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed overall, small number of patients completing questionnaire in the control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03296566/ICF_000.pdf
  • Study Protocol (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03296566/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT03296566/SAP_002.pdf